CLINICAL TRIAL: NCT06373952
Title: Integrated Online-to-offline (O2O) Model of Care for HIV Prevention and Treatment Among Men Who Have Sex with Men
Acronym: CINTAI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, Roman Shrestha, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-08-658-910
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: HIV Prevention Program
Keywords: HIV; men who have sex with men; website
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CINTAI (Experimental): Participants randomized to the Jom-TestPlus group will have access to all Jom-TestPlus features, including: assessment center; online registration; risk calculator; HIVST kit order, management, and monitoring; automated reminders; real-time e-counseling (eHIVST, active referral services); chemsex-related harm reduction services (screening, chemsex e-counseling, PartyPack ordering), chat function (ability to chat with counselors and research staff); and knowledge center (multimedia library on information and resources on HIV testing, PrEP, treatment, risks, and chemsex). Participants will follow a defined pathway to accessing HIVST kit ordering, e-counseling, and subsequent O2O linkage to clinical services.
  Interventions: Behavioral: Online to offline counseling
- Control (Active Comparator): being deactivated. The TAU group will have access to the assessment center (risk assessment, follow-up surveys), knowledge center (multimedia library on information and resources on HIV testing, PrEP, treatment, risks, and chemsex), and a voucher for no-cost community-based HIV testing (sent via secure, encrypted email or can be downloaded on the Jom-TestPlus).
  Interventions: Behavioral: Online to offline counseling

INTERVENTIONS:
Behavioral: Online to offline counseling — * Online registration and risk assessment: Users complete an onboarding process comprised of creating an account, entering demographic data, customizing settings, and completing the baseline risk assessment.
  * HIVST kit order, management, and monitoring: The platform will allow users to request HIVST kits via standard mail or self-pickup at user-preferred sites (e.g., LGBT-friendly clinics). After completing the mandatory section of the questionnaire and selecting a delivery option, a random personal identification number will be assigned by the system, which will be used to track future HIVST requests, collect HIVST results, and monitor subsequent linkage to further testing and HIV care.
  * eHIVST and O2O linkage to HIV clinical services: After unsealing the test kit, participants will find a reminder card to schedule their O2O pre- and post-test e-counseling appointment.

SUMMARY:
The proposed research focuses on developing and testing a web-based platform, called Jom-TestPlus, that will incorporate HIV self-testing (HIVST) with real-time e-counseling (eHIVST) with online-to-offline (O2O) linkage to HIV prevention and treatment services while simultaneously co-addressing chemsex-related needs for men who have sex with men (MSM) in Malaysia. This model represents a potentially impactful strategy for reaching marginalized populations, like MSM, and allows immediate engagement in the post-test linkage process to prevention or treatment services.

DETAILED DESCRIPTION:
Malaysia's HIV epidemic is rapidly expanding, with recent evidence suggesting increasing sexual transmission, especially in MSM. HIV prevalence among MSM is now at an all-time high of 21.6% and is concentrated in the country's capital, Kuala Lumpur, where prevalence among MSM is 43% in 2020, up from 22% just four years before. Insights into Malaysia's expanding HIV epidemic are multi-factorial: Both homosexuality and substance use are criminalized in Malaysia. MSM are, therefore, often hesitant to disclose their sexuality or risk behaviors, primarily due to fear of stigma, discrimination, or criminalization. Further, evidence suggests the widespread use (24%) of psychoactive substances (e.g., amphetamine-type stimulants) before or during a sexual encounter, also known as sexualized drug use (chemsex) among Malaysian MSM, which leads to high-risk sexual practices (e.g., condomless sex). Stigma and discrimination are also enacted on MSM by healthcare providers, which foster a hostile environment toward MSM, complicating efforts to scale-up of HIV testing and subsequent linkage to HIV prevention (pre-exposure prophylaxis) and treatment (antiretroviral therapy) services. HIV testing jumpstarts entry into the HIV prevention and treatment cascades. New HIV testing guidelines recommend MSM test every 3 to 6 months, as early HIV testing is a cost-effective strategy for stemming the HIV epidemic. Yet, HIV testing rates remain low among Malaysian MSM: ever tested (70.3%) and last year tested (30.9%). HIV selftesting (HIVST) may be particularly impactful among MSM in Malaysia. Although willingness to use HIVST is high in this group, its use is still minimal due to lack of access to HIVST kits, concerns related to misinterpreting results, and missed opportunities for counseling and linkage to care. In this context, eHealth represents an innovative platform to transform the face of HIV service delivery (i.e., testing and linkage to care). Leveraging eHealth platforms for HIV services delivery in Malaysia is ideal given that nearly all (>99%) MSM use some form of communication technology (e.g., smartphone, laptop) and has a strong preference for web-based platforms for HIVST. Therefore, a web-based HIVST platform, called Jom-Test®, was developed to promote HIV testing by providing free anonymous HIVST. The results demonstrated high feasibility and acceptability for the platform but low post-test linkage to treatment and prevention services. The findings further indicated the need for real-time (online) access to counselors for pre- and post-test counseling and support for linkage to HIV and chemsex-related harm reduction services (offline). To address this evidence gap, this application proposes to jump-start the broader HIV care continuum by adapting, expanding, and refining an existing Jom-Test® platform. The enhanced version, to be called Jom-TestPlus, will include real-time e-counseling (eHIVST) with integrated O2O linkage to HIV prevention and treatment services while simultaneously co-addressing chemsex-related needs for Malaysian MSM. This model represents a potentially impactful strategy for reaching marginalized populations, like MSM, and allows immediate engagement in the post-test linkage process to prevention or treatment services.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥18 years;

  * Cisgender male;
  * HIV-negative or HIV status unknown;
  * Own or have access to a computer, tablet, or internet-enabled smartphone

Exclusion Criteria:

* • Unable to provide informed consent

  * Unable to read and understand English or Bahasa Malaysia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
HIVST uptake | Time Frame: 3 and 6 months post-randomization
  Uptake of HIV self-testing (yes/no) will be assessed at each follow-up time point (3 and 6 months) using self-reported measure.
Linkage to PrEP | Time Frame: 3 and 6 months post-randomization
  Linked to PrEP services (yes/no) will be assessed at each follow-up time point (3 and 6 months) using self-reported measure.
Linkage to HIV treatment services | Time Frame: 3 and 6 months post-randomization
  Linked to ART services (yes/no) will be assessed at each follow-up time point (3 and 6 months) using self-reported measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Excellence For Research in AIDS (CERiA), Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No